CLINICAL TRIAL: NCT02331810
Title: A Randomized, Double-blind, Placebo-controlled Study Of Safety, Tolerability, And Pharmacokinetics Of Repeated Ascending Subcutaneous Doses Of SAR113244 And Pharmacodynamics Of Single Dose Of SAR113244 In Male And Female Lupus Patient
Brief Title: Pharmacodynamics Assessment Study After Single Subcutaneous Dose Of SAR113244 Versus Placebo In Lupus Male And Female Patients
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PDY14076; 2014-001690-13 (EudraCT Number); U1111-1154-6184 (Other: UTN)
Record Dates: First submitted 2014-12-05; First posted 2015-01-06 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SAR113244 (Experimental): Single subcutaneous dose of SAR113244
  Interventions: Drug: SAR113244
- Placebo (Placebo Comparator): Single subcutaneous dose of placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: SAR113244 — Pharmaceutical form:solution for injection Route of administration: subcutaneous
  Arms: SAR113244
Drug: placebo — Pharmaceutical form:solution for injection Route of administration: subcutaneous
  Arms: Placebo

SUMMARY:
Primary Objective:

Assess in systemic lupus erythematosus (SLE) patients the effect of SAR113244 on B-cell subsets compared to placebo.

Secondary Objectives:

Assess in male and female lupus patients after SC single dose of SAR113244 the tolerability and safety of SAR113244.

Assess in male and female lupus patients:

* The pharmacokinetics of SAR113244.
* The pharmacodynamics of SAR113244 for the following disease parameters:

  * Safety of Estrogens in Lupus Erythematosus National Assessment Systemic Lupus Erythematosus Disease Activity Index (SELENA-SLEDAI) score, British Isles Lupus Assessment Group (BILAG) score (if applicable), BILAG-Based Composite Lupus Assessment (BICLA) (if applicable), systemic lupus erythematosus responder index (if applicable), Lupus-quality of life and Functional Assessment of Chronic Illness Therapy-Fatigue, anti-double stranded deoxyribonucleic acid antibody and anti-nuclear antibody levels and plasma complement levels (C3, C4), erythrocyte sedimentation rate and C-reactive protein.
  * Peripheral blood B and T cell subsets.

DETAILED DESCRIPTION:
The total duration of screening to end of study per subject is 16 weeks with post-study observation on Day 198 for anti-drug antibody assessment (for patients with positive anti-drug antibody at end of study only).

ELIGIBILITY:
Inclusion criteria:

* Male or female patients, between 18 and 75 years of age, inclusive.
* Clinical diagnosis of SLE by American College of Rheumatology (ACR) criteria.
* Autoantibody-positive.
* On active and stable SLE disease.
* B cell subsets expressed as percentage of total B cells above normal.

Exclusion criteria:

* Pregnant and nursing.
* Have received treatment with investigational drugs in the 4 months prior to the screening or 5 half-lives of the drug, which ever is longer.
* Have received intravenous or oral cyclophosphamide within 180 days of Day 0.
* Severe active lupus nephritis or chronic renal insufficiency.
* Active or chronic, severe neuropsychiatric lupus.
* Acute, recent (within 4 weeks of screening), chronic or frequently recurring infection(s), except minor infection.
* Have current drug or alcohol abuse or dependence.
* Have a historically positive test or test positive at screening for HIV, hepatitis B, or hepatitis C.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Percentage decrease in B cell subsets (expressed as percentages of total B-cells) from baseline | Up to Day 57 after inclusion

SECONDARY OUTCOMES:
Assessment of pharmacokinetic parameter - maximum concentration (Cmax) | Up to Day 198 after inclusion
Assessment of pharmacokinetic parameter - time of maximum concentration (Tmax) | Up to D198 after inclusion
Assessment of pharmacokinetic parameter - area under curve from zero to infinity (AUCinf) | Up to Day 198 after inclusion
Assessment of pharmacokinetic parameter - time of the last point with quantifiable concentration (tlast) and terminal elimination half-life (t1/2z) | Up to Day 85 after inclusion
Assessment of pharmacokinetic parameter-apparent oral clearance (CL/F) | Up to Day 85 after inclusion
Assessment of pharmacokinetic parameter- absorption-dependent apparent volume of distribution at steady state (Vss/F) | Up to Day 85 after inclusion
Number of participants with anti-SAR113244 antibody titers | Up to Day 198 after inclusion
Number of participants with adverse events and treatment-emergent adverse events, including those that deviated from baseline values of hematology, biochemistry, coagulation and urine | Up to Day 198 after inclusion
Number of participants with injection site reactions | Up to Day 85 after inclusion
Number of participants with abnormalities and changes in laboratory parameters | Up to Day 85 after inclusion
Assessment of pharmacodynamics - clinical and/or lupus-related scores | Up to Day 85 after inclusion
Assessment of pharmacodynamics - blood/urine parameters | Up to Day 85 after inclusion
Pharmacodynamic parameters: peripheral blood B and T cells subsets | Up to Day 85 after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi